CLINICAL TRIAL: NCT06473792
Title: Effect of Probiotic Toothpaste and Regular Toothpaste on Plaque Levels of Orthodontic - A Randomized Controlled Trial
Brief Title: Effect of Probiotic Toothpaste and Regular Toothpaste on Plaque Levels of Orthodontic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanza Tahir (Other)
Responsible Party: Sponsor-Investigator, Kanza Tahir, Dr. Kanza Tahir, Aga Khan University
Organization: Aga Khan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-7853-26493
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Plaque
Keywords: Plaque; Gingivitis; Probiotics
MeSH Terms: conditions — Plaque, Amyloid; Gingivitis

STUDY DESIGN:
Masking Description: For reexamination at T1, the investigators were blinded to the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colgate Maximum Cavity Protection (Control) (No Intervention): Participants will be advised to use regular toothpaste twice a day for 3 weeks after the bonding. A regular toothpaste and a standard brushing technique will be conveyed to all the participants.
- Probiotic Toothpaste Group (Experimental): Participants will be advised to use a Probiotic toothpaste twice a day for 3 weeks after the bonding. A probiotic toothpaste and a standard brushing technique will be conveyed to all the participants.
  Interventions: Other: Probiotic Toothpaste

INTERVENTIONS:
Other: Probiotic Toothpaste — Composition: Main - Water, calcium carbonate, calcium glycerophosphate, glycerin, xylitol, sodium bicarbonate, sweet fennel oil (Foeniculum vulgare), carrageenan, maltodextrin, Dental-Lac (Lactobacillus paracasei), potassium sorbate, yucca (Y. filamentosa) powder, stevia leaf extract (Eupatorium rebaudiana bertoni), zinc chloride.
  Usage: This is mint flavored toothpaste containing Lactobacillus paracasei which has demonstrated the ability to help address harmful strains of oral flora, and promotes the maintenance of a healthy teeth and gums. The participant will be instructed to brush with it twice daily.
  Other Names: PerioBiotic Toothpaste - Dental Probiotic Tooth Paste
  Arms: Probiotic Toothpaste Group

SUMMARY:
This study is set to determine the improvement in plaque levels utilizing Plaque Index Simplified scores in orthodontic patients using probiotic toothpaste and regular toothpaste.

It will further analyze the mean difference in oral hygiene scores between metal and ceramic brackets in regular toothpaste and probiotic toothpaste groups.

DETAILED DESCRIPTION:
Probiotic toothpaste is formulated to introduce beneficial bacteria into the oral cavity, promoting a balanced microbiome and inhibiting the growth of pathogenic bacteria. Previous research suggests that probiotics can reduce plaque formation, gingival inflammation, and pathogenic bacterial load. By potentially improving the oral microbiome, probiotic toothpaste could offer a superior alternative to standard toothpaste for maintaining oral hygiene in orthodontic patients. Metal and ceramic brackets differ not only in aesthetics but also in their interaction with the oral environment. Ceramic brackets are more brittle and can be more prone to plaque accumulation due to their rougher surface compared to metal brackets. This study will determine the improvement in plaque levels utilizing Plaque Index Simplified scores in orthodontic patients using probiotic toothpaste and regular toothpaste.

It will further determine the mean difference in oral hygiene scores between metal and ceramic brackets in regular toothpaste and probiotic toothpaste groups.

Plaque will be assessed using plaque disclosing tablets before the bonding (T1) and 3 weeks after the bonding (T2). The data will be collected on Plaque Index Simplified chart. Eligible participants will be randomly allocated to one of the two groups.

Group A (Control): Participants will be advised to use regular toothpaste twice a day for 3 weeks after the bonding. A standard toothpaste and brushing technique will be conveyed to all the participants.

Group B (Intervention): Participants will be advised to use a Probiotic toothpaste twice a day for 3 weeks after the bonding. A probiotic toothpaste and brushing technique will be conveyed to all the participants.

The total sample size for each group would be 26. Since this study has 2 groups, a total number of 52 (N) will be required. Group 1: Regular toothpaste and Group 2: Probiotic toothpaste.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will be initiating their orthodontic treatment by bonding of metal or ceramic brackets
* Patients age between 18 - 50 years
* Patients without any mental and physical disability or craniofacial disorders
* Patients without enamel or dentin dysplasia
* Patients not taking medications affecting plaque accumulation such as antibiotics or antibacterial mouth rinses
* Patients without periodontal disease or dental caries at the study onset
* Patients willing to follow-up after 3 weeks

Exclusion Criteria:

* Patients with neurological mental deficits or otherwise medically compromised
* Patients with past history of dental trauma or craniofacial syndromes
* Patients who are smokers
* Those patients who are already continuing their orthodontic treatment
* Patients with poor oral hygiene

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2024-06-04 (Actual); Primary Completion 2024-07-06 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Plaque Index Simplified | Before and three weeks after bonding
  Number of sites with plaque/ Number of sites evaluated x 100
Gingival Index | Before and three weeks after bonding
  Gingival Index measures gingival condition of the marginal and interproximal tissues (mesial, lingual, distal, facial) separately on the basis of 0 to 3 with 0=Normal gingiva; 1= Mild inflammation - slight change in color and slight edema but no bleeding on probing; 2= Moderate inflammation - redness, edema and glazing, bleeding on probing; 3= Severe inflammation - marked redness and edema, ulceration with tendency to spontaneous bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Mubassar Fida, FCPS, MCPS, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tahir K, Barakaat AA, Shoukat Ali U, Fida M, Sukhia RH. Effect of probiotic toothpaste and regular toothpaste on gingival health and plaque levels of adult orthodontic patients - An open label randomized controlled trial. Int Orthod. 2025 Mar;23(1):100938. doi: 10.1016/j.ortho.2024.100938. Epub 2024 Oct 30. PMID 39476739